CLINICAL TRIAL: NCT06060808
Title: Role of NFKBIA and PTPN22 Genes Polymorphism in Acute Rejection Susceptibility After Living Donor Liver Transplantation in Egyptian Patients.
Status: Completed | Type: Observational
Sponsor: Helwan University (Other)
Responsible Party: Principal Investigator, Sara Mohamed Mohamed Abdel Motaleb, lecturer, Helwan University
Other Study IDs: gene polymorphism
Record Dates: First submitted 2023-09-24; First posted 2023-09-29 (Actual); Last update posted 2023-09-29 (Actual); Status verified 2023-09

CONDITIONS: Liver Transplant Rejection
Keywords: gene polymorphism
MeSH Terms: interventions — Polymorphism, Genetic

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 2 Years
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Genetic: gene polymorphism — gene polymorphism of NFKBIA and PTPN22 genes

SUMMARY:
Our study aimed at studying the impact of gene polymorphism of NFKBIA and PTPN22 genes on rejection episodes in liver transplant Egyptian recipients. Also assess patients' factors associated with graft rejection.

DETAILED DESCRIPTION:
Liver transplantation is considered an effective therapy for severe liver disease, but graft dysfunction occurs in up to 13% of patients during the first year following transplantation, and rises to 35% after 5 years (Keeffe, 1999; Yu et al., 2001). Graft rejection is one of the major immunological complications following liver transplantation (Zheng et al., 2006).

The nuclear factor of kappa light polypeptide gene enhancer B-cells inhibitor-alpha (NFKBIA) gene encodes a member of the nuclear factor-kappa-B inhibitor family. Polymorphisms in this gene might be associated with a susceptibility to acute rejection episodes following liver transplantation, as they may cause an increased activation level of the proinflammatory transcription factor nuclear factor of kappa light polypeptide gene enhancer in B-cells (NFκB).

NFκB translocates to the nucleus and promotes the expression of a panel of genes (Karin and Ben-Neriah, 2000). Some of these, for example interleukin-2, interleukin-6, interleukin-12 or tumor necrosis factor-alpha, play an important role in the pathogenesis of allograft rejection and the activation of the immune system in general (Wei and Zheng, 2003).

The protein tyrosine phosphatase nonreceptor 22 gene (PTPN22) encodes a strong T-cell regulator called lymphoid protein tyrosine phosphatase. Previously, PTPN22 was described as a susceptibility gene for autoimmunity because it contains single nucleotide polymorphisms (SNPs) associated with several autoimmune diseases. One SNP (rs2476601;1858G>A) has emerged as a particularly potent risk factor for autoimmunity. We address the question whether PTPN22 polymorphismsare also associated with acute rejection after liver transplantation. (Dullin et al., 2015).

ELIGIBILITY:
Inclusion Criteria:

* Adult Patients with ESLD were subjected to living donor liver transplantation due to different etiologies including hepatitis C virus (HCV), hepatitis B virus (HBV), autoimmune hepatitis (AIH), portal venous thrombosis (PVT), cryptogenic hepatitis, Primary sclerosing cholangitis(PSC), hepatocellular and carcinoma(HCC) were eligible for the study. Recipients received calcineurin inhibitors either tacrolimus or cyclosporine as primary immunosuppressant ± MMF or evorilumus ± MMF immediately after transplantation.

Exclusion Criteria:

* Patients were excluded if they had multi-organ transplantation, had previously received a liver transplant, or were receiving an ABO-incompatible transplant.

Ages: 20 Years to 64 Years | Sex: All
Age Groups: Adult
Study Population: Adult patients with end stage liver disease(ESLD) underwent living donor liver transplantation were recruited from Ain Shams University hospitals, Cairo, Egypt.
Sampling Method: Non-Probability Sample
Enrollment: 105 (Actual)
Dates: Start 2021-03-15 (Actual); Primary Completion 2023-04-23 (Actual); Study Completion 2023-07-24 (Actual)

PRIMARY OUTCOMES:
gene polymorphism | baseline
  gene polymorphism of NFKBIA and PTPN22 genes

SECONDARY OUTCOMES:
immunosuppressant levels | 14 days
  tacrolimus,cycosporin,evrolimus trough levels

CONTACTS AND LOCATIONS:
Locations (1):
- Sara Mohamed Mohamed, Cairo, Egypt